CLINICAL TRIAL: NCT00804700
Title: Impact of Two Methods of Listening to Music During Exercise on Perceived Exertion and Overall Physical Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Responsible Party: Rebecca Over, DO, Georgetown University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2008-316
Record Dates: First submitted 2008-12-08; First posted 2008-12-09 (Estimated); Last update posted 2010-04-23 (Estimated); Status verified 2008-12

CONDITIONS: Sedentary Lifestyle
Keywords: synchronous; exercise; music; heartbeat; tunes
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (Active Comparator): Subjects will be given a 60 minute lecture on the benefits of regular exercise and how music can enhance the exercise experience. Subjects will be individually instructed how to use the Precor elliptical trainer at the Yates fitness center while listening to music. Subjects are instructed to exercise using the elliptical trainer for periods of 45 -55 minutes at a time as frequently as they like with a minimum frequency of once per week. Subjects will also be encouraged to exercise regularly by walking, jogging or engaging in other forms of physical activity during the intervention period. A fitness attendant will be on hand to supervise their exercise activity, but will not give specific advice how to exercise, other than to make sure they are exercising safely.
  Interventions: Behavioral: Active teaching in synchronous listening to music while exercising
- Intervention Arm (Experimental): Subjects will be instructed to exercise while listening to four audio tutorials that are stored on their MP-3 player. These tutorials guide the subject on how to synchronize his or her body movements to the beat of the music.
  Interventions: Behavioral: Active teaching in synchronous listening to music while exercising

INTERVENTIONS:
Behavioral: Active teaching in synchronous listening to music while exercising — Subjects will be instructed to exercise while listening to four audio tutorials that are stored on their MP-3 player. These tutorials guide the subject on how to synchronize his or her body movements to the beat of the music.

SUMMARY:
The purpose of the study is to compare two different methods of listening to music while performing aerobic exercise: synchronous music listening vs. asynchronous music listening. Synchronous music listening while exercising is a learned activity where the participant moves his or her body in synchrony with the beat of the music, similar to dancing or to participating in a group exercise (aerobics) class. Our hypothesis is that synchronous music listening reduces the level of perceived exertion to the exercise and motivates the subject to exercise more often. This study randomly assigns 46 subjects, age 20-55 years old to either a control group of listening to their own favorite music in an asynchronous fashion or to an intervention group of listening to prepared music in a synchronous fashion over a six week period.

ELIGIBILITY:
Inclusion Criteria:

* Adult employees of Georgetown University (age 20-55) who listen to music while exercising.

Exclusion Criteria::

* A major medical condition that would prevent the participant from undertaking regular exercise
* The use of beta blocker medication
* Participation in varsity sports

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2008-12; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Change in Borg Rating of Perceived Exertion (RPE) from baseline to final test at 6 weeks intervention | 6 weeks

SECONDARY OUTCOMES:
Difference in exercise-related energy expenditure over six weeks between to intervention and control groups | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Georgetown University, Washington D.C., District of Columbia, United States